CLINICAL TRIAL: NCT04127136
Title: Effects of Multi-Disciplinary Training Therapy On Binge Eating Episodes
Brief Title: Analysis of the Effects of the Adana City Training and Research Hospital Obesity Center Training Program on Adult Obese Patients With Binge Eating Disorder. A Prospective, Quasi-experimental Study With Interrupted Time-series Design.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Cenk Belibağlı, Obesity Center Manager, Family Physician, Adana City Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 483
Record Dates: First submitted 2019-10-14; First posted 2019-10-15 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Binge-Eating Disorder; Group Meetings; Weight Loss
Keywords: obesity; weight loss; Binge-Eating Disorder
MeSH Terms: conditions — Obesity; Binge-Eating Disorder; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): The cases were analyzed for the change in the severity of binge eating disorder in the program. The data collection was performed via socio-demographic information form, binge eating disorder evaluation (BEDE) form, and progress record forms. BEDE was a structured form exclusively using DSM-5 BED diagnosis and the severity criteria. Progress record form included weekly session content that was administered by a physician, dietitian, psychologist, and the physiotherapist and the monthly individual meetings data. BEDE and progress record forms were applied before the trainings that focuses on cognitive change and repeated every four weeks for 20 weeks. The patients were planned to receive 80 hours of training by the physician, dietitian, psychologist, and the physiotherapist.
  Interventions: Behavioral: Multi-disciplinary obesity management therapy

INTERVENTIONS:
Behavioral: Multi-disciplinary obesity management therapy — In twenty weeks, trainings by the physician, dietitian, psychologist and physiotherapist are conducted about medical information about obesity, using the technology to aid weight loss, what, when, how and why to eat, nutrition groups, ration management, water consumption, self-awareness, stress management, obesity and the association between the psychological processes, warming up and mobilization, correct stance and posture, and adequate physical activity. In addition to group meetings, in monthly individual meetings, the progress of the patients are evaluated.

SUMMARY:
Outcomes of treatments for binge eating spectrum eating disorders are yet to yield desirable results, reporting up to 60-70% of patients remaining symptomatic at post-treatment.

Adana City Training and Research Hospital Obesity Center is designed to provide multi-disciplinary health care services and training for groups of obese patients seeking professional help. The center includes a physician, dietitian, physiotherapist, psychologist, public relations officer, and a nurse acting as a life coach. Program is planned to carry initial assessment, health screening, necessary medical attention related to obesity, cognitive change, behavioral change, and sustainability activities. The initial assessment part consisted of one on one interviews of the patient with the physician, psychologist, dietitian, physiotherapist, and the nurse. Then, the patient is consulted with an endocrinologist, cardiologist, psychiatrist, and physical therapy and rehabilitation specialist to elucidate the significant factors that resulted in excessive weight gain and barriers in losing. Patients with severe or mismanaged medical conditions, including chronic diseases, neurological diseases, significant affective and psychotic disorders, and substance abuse or addiction disorders were directed to relevant clinics before registration. The patients who completed the screening are arranged into groups and weekly group meetings are planned. In two group meetings, basic medical knowledge and frequently asked questions are discussed. The center staff and the patients get acquinted. In the following twenty weeks, trainings by the physician, dietitian, psychologist and physiotherapist are conducted about medical information about obesity, using the technology to aid weight loss, what, when, how and why to eat, nutrition groups, ration management, water consumption, self-awareness, stress management, obesity and the association between the psychological processes, warming up and mobilization, correct stance and posture, and adequate physical activity. In addition to group meetings, in monthly individual meetings, the progress of the patients are evaluated.

During the course of the program the patients with BED reported improvements in BED episodes and increased weight loss rate which give the idea to conduct a study. The primary goal of the study was to analyze the change in the severity of binge eating disorder in patients registered to the program. We expected to show a decrease in the frequency of the BED episodes in all the patients. The secondary goal includes the analysis of the context of the training program to compare the effectiveness of the topics and the methods.

The study was a single-arm, prospective, quasi-experimental study with interrupted time-series design. There were no sampling methods; all patients registered to the center program with binge eating disorder and completed the acquaintance step were asked to be included. Inclusion criteria were having registered to the center for training, passed the first three steps, age between 18 to 65 years, a body mass index (BMI) equal to or over 30, and having binge eating disorder. Patients who failed to attend more than four pieces of training and complete a binge eating evaluation were excluded from the study. The training materials were developed by the trainers and edited by the author for the final version before training.

The cases were analyzed for the change in the severity of binge eating disorder in the program. The data collection was performed via socio-demographic information form, binge eating disorder evaluation (BEDE) form, and progress record forms. BEDE was a structured form exclusively using DSM-5 BED diagnosis and the severity criteria1. Progress record form included weekly session content that was administered by a physician, dietitian, psychologist, and the physiotherapist and the monthly individual meetings data. BEDE and progress record forms were applied before the trainings that focuses on cognitive change and repeated every four weeks for 20 weeks. The patients were planned to receive 80 hours of training by the physician, dietitian, psychologist, and the physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* having registered to the center for training
* passed the first three steps
* body mass index (BMI) equal to or over 30
* having binge eating disorder

Exclusion Criteria:

* having an untreated medical condition
* having a mismanaged medical condition
* failing to attend more than 4 meetings
* failing to complete a binge eating disorder evaluation form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Change in the severity of binge-eating disorder | 20 weeks
  The Binge eating disorder form, constructed exclusively using DSM-5 BED diagnosis and the severity criteria, was consisted of 12 questions, addressing major criteria including the characterization of recurrent episodes of binge eating and the sense of lack of control over eating during the episode, the feelings at the time and after eating, the presence of distress and finally the frequency. Based on the frequency of episodes, four severity groups were set according to the weekly episodes: mild, moderate, severe, and extreme, respectively. The first ten questions were in closed forms and designed to detect the presence or the characterization of the episodes. Answers with "yes" reflect the presence of the symptoms or the episodes and mean a worse outcome. The last two focus on the frequency of the symptoms. Higher scores mean a worse outcome. We expected the subjects to show a change in the severity of binge eating episodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Training and Research Hospital Obesity Center, Yüreğir, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qian J, Hu Q, Wan Y, Li T, Wu M, Ren Z, Yu D. Prevalence of eating disorders in the general population: a systematic review. Shanghai Arch Psychiatry. 2013 Aug;25(4):212-23. doi: 10.3969/j.issn.1002-0829.2013.04.003. PMID 24991159
- [Background] Bulik CM, Kleiman SC, Yilmaz Z. Genetic epidemiology of eating disorders. Curr Opin Psychiatry. 2016 Nov;29(6):383-8. doi: 10.1097/YCO.0000000000000275. PMID 27532941
- [Background] Dakanalis A, Riva G, Serino S, Colmegna F, Clerici M. Classifying Adults with Binge Eating Disorder Based on Severity Levels. Eur Eat Disord Rev. 2017 Jul;25(4):268-274. doi: 10.1002/erv.2518. Epub 2017 Apr 20. PMID 28425618
- [Background] Linardon J. Meta-analysis of the effects of cognitive-behavioral therapy on the core eating disorder maintaining mechanisms: implications for mechanisms of therapeutic change. Cogn Behav Ther. 2018 Mar;47(2):107-125. doi: 10.1080/16506073.2018.1427785. Epub 2018 Jan 30. PMID 29378481
- [Background] Sedgwick P, Greenwood N. Understanding the Hawthorne effect. BMJ. 2015 Sep 4;351:h4672. doi: 10.1136/bmj.h4672. No abstract available. PMID 26341898